CLINICAL TRIAL: NCT01112514
Title: A Pilot Study of Indocyanine Green Fluorescent Molecular Imaging of the Gastrointestinal Tract
Brief Title: Indocyanine Green Fluorescent Molecular Imaging of the Gastrointestinal Tract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); National Cancer Institute (NCI) (NIH); Damon Runyon Cancer Research Foundation (Other)
Responsible Party: Principal Investigator, Andrew T. Chan, MD, MPH, Study Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-398
Record Dates: First submitted 2010-04-27; First posted 2010-04-28 (Estimated); Results first posted 2014-02-24 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-01

CONDITIONS: High Risk Polyposis Syndrome; Distal Colonic Lesions; Colorectal Polyps
Keywords: ICG; indocyanine green
MeSH Terms: interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ICG Injection (Experimental): These participants underwent a colonoscopy after having an ICG injection.
  Interventions: Drug: indocyanine green

INTERVENTIONS:
Drug: indocyanine green — Administered intravenously during endoscopic near-infrared (NIR) imaging
  Other Names: ICG; IC-Green

SUMMARY:
Standard white light endoscopy involves the passage of a thin, flexible camera into the colon from the anus. Although standard white light endoscopy can detect most polyps and precancerous areas in the gastrointestinal tract and colon, many studies have shown that even the most experienced doctors, under optimal conditions, can miss up to 15-25% of precancerous areas. Thus, there remains a clear need to develop new methods of improving standard white light endoscopy. We are investigating whether indocyanine green (ICG) can serve to highlight areas which are precancerous when the colon is visualized with a special cameral which shines fluorescent light. Information from other studies suggests that this ICG agent may help to visualize blood vessels flowing to precancerous areas in the colon. We are looking at the ability of ICG, in combination with an endoscope which shines fluorescent light, to visualize precancerous areas in the colon.

DETAILED DESCRIPTION:
* Participants will be scheduled for their regular lower endoscopy. On the day of the procedure, participants will come to the endoscopy unit at Massachusetts General Hospital. After arriving, participants will receive an intravenous line and meet with the research doctor to go over the procedure. The participant will then be transferred to the endoscopy procedure room and be administered sedatives until they are comfortable to proceed with the procedure.
* The research doctor will pass the flexible study sigmoidoscope into the lower part of the rectum. At this time, a dose of the ICG contrast agent will be administered through the intravenous line. Any areas that are suspicious will be photographed using the camera in the scope. We will also biopsy/remove any suspicious areas and send it to the pathologist as we normally do during endoscopy.
* Over the course of the study procedure, small doses of ICG will be administered to help find any precancerous areas. Altogether, the study exam should not take more than 10 to 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Participants will include patients with high risk polyposis syndromes with planned routine endoscopic surveillance for neoplasia or patients with planned endoscopic evaluation of distal colonic lesions suspicious for colorectal polyps or cancer detected on abdominal imaging
* Fit for conscious sedation or monitored anesthesia care for colonoscopy-American Society of Anesthesiologists (ASA) Class I or II
* 18 years of age or older
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-2
* Negative human chorionic gonadotropin (HCG) test for women of child-bearing age. Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation

Exclusion Criteria:

* Participants with AsA class III, IV, V
* Documented allergy to iodine, iodine-containing compounds of ICG
* Documented allergy to sulfur containing compounds
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ICG
* History of adverse reactions to endoscopy or sedatives for endoscopy
* Pregnant or breast-feeding women
* Participants who are unable to discontinue warfarin anticoagulation 5 days before the procedure
* Participants taking phenobarbital, phenylbutazone, primidone, phenytoin, haloperidol, nitrofurantoin, probenecid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T. Chan, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four participants were enrolled in the study, and of these four, one withdrew from the study. All participants were recruited between April 2010 and May 2012.
Groups:
- ICG Injection: Participants received an Indocyanine Green Fluorescent (ICG) injection in order to study imaging of the colon during a colonoscopy.
Period: Overall Study
Arm/Group | ICG Injection
Started | 4
Completed | 3
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: One participant withdrew from the study.
Arm/Group | ICG Injection
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (9.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Neoplastic Lesions Detected
Time Frame: upto 15 mins
Measure: Number; unit: Lesions
Arm/Group | ICG Injection
Number analyzed (Participants) | 3
Lesions | 3

ADVERSE EVENTS:
Arm/Group | ICG Injection
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No